CLINICAL TRIAL: NCT06409429
Title: A Prospective, Multicenter, Randomized, Double-blind, Placebo-controlled Study of Nimotuzumab Combined With GX as Postoperative Adjuvant Therapy in Pancreatic Cancer
Brief Title: Nimotuzumab Combined With GX as Postoperative Adjuvant Therapy in Pancreatic Cancer
Status: Not yet recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Tianjin Medical University Cancer Institute and Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IST-Nim-PC-45
Record Dates: First submitted 2024-05-07; First posted 2024-05-10 (Actual); Last update posted 2024-05-10 (Actual); Status verified 2024-05

CONDITIONS: Pancreatic Cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — nimotuzumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Nimotuzumab+ GX) (Experimental)
  Interventions: Drug: Nimotuzumab; Drug: GX
- Control group (Placebo+ GX) (Placebo Comparator)
  Interventions: Drug: GX; Drug: Placebo

INTERVENTIONS:
Drug: Nimotuzumab — Patients will receive Nimotuzumab 400 mg weekly or Nimotuzumab 600 mg on Day 1 and 8 of a 21-day cycle, up to 6 months.
  Other Names: h-R3
  Arms: Experimental group (Nimotuzumab+ GX)
Drug: GX — Patients will receive GX as adjuvant therapy for 6 months. Gemcitabine will be delivered as a 1000 mg/m² intravenous infusion administered on Day 1 and 8 of a 21-day cycle. Capecitabine 2000mg/m²/day will be administered orally for 14 days followed by 7 days' rest.
Drug: Placebo — Patients will receive placebo 400 mg weekly or placebo 600 mg on Day 1 and 8 of a 21-day cycle, up to 6 months.
  Arms: Control group (Placebo+ GX)

SUMMARY:
This is a prospective, multicenter, randomized, double-blind, placebo-controlled study. The main purpose of the study is to evaluate the clinical efficacy and safety of Nimotuzumab combined with GX for postoperative adjuvant treatment of pancreatic cancer.

DETAILED DESCRIPTION:
This clinical study is designed as a prospective, multicenter, randomized, double-blind, placebo-controlled study to evaluate the clinical efficacy and safety of Nimotuzumab combined with GX (gemcitabine plus capecitabine) compared with GX only for resected pancreatic cancer. About 146 patients will be enrolled in this study and randomly divided into experimental group (nimotuzumab plus GX) and control group (placebo plus GX) at a ratio of 1:1. The main endpoint is relapse-free survival (RFS). Additional end points included distant metastasis-free survival (DMFS), overall survival (OS), tumor-related markers and safety.

ELIGIBILITY:
Inclusion Criteria:

* 1. Able and willing to provide a written informed consent.
* 2. Age 18-75 years old, gender unlimited;
* 3. Histologically or cytologically confirmed resected pancreatic ductal adenocarcinoma (PDAC), resectable evaluation is based on criteria of NCCN guidelines, no evidence of distant metastasis as demonstrated by imaging;
* 4. Postoperative pathology suggested R0/R1 resection;
* 5. Adequate organ and bone marrow function, defined as follows: absolute neutrophil count (ANC)≥1.5×10^9/L; platelets≥100×10^9/L; hemoglobin≥9.0 g/dL; serum total bilirubin (TBIL)≤1.5×ULN; aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 2.5 times the upper limit of normal (ULN); serum creatinine≤1.5×ULN or estimated creatinine clearance > 60 mL/min;
* 6. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1;
* 7. Postoperative survival is expected to be ≥3 months;
* 8. Fertile subjects are willing to take contraceptive measures during the study period.

Exclusion Criteria:

* 1. Prior neo-adjuvant treatment, radiation therapy, or systemic therapy for pancreatic adenocarcinoma;
* 2. Accompanied by other serious diseases, including but not limited to: active infections; unmanageable diabetes mellitus and uncontrolled hypertension (SBP>160mmHg or DBP>100mmHg); compensatory heart failure (NYHA grade III and IV), unstable angina or poorly controlled arrhythmias within 3 months prior to randomization; presence of uncontrolled pleural effusion, pericardial effusion, or ascites requiring drainage; severe portal hypertension; gastric outlet obstruction; Respiratory insufficiency and Severe lung disease; Central Nervous System Disease or mental illness;
* 3. History of other malignancies (except cured basal cell carcinoma of the skin and carcinoma in situ of the cervix);
* 4. bleeding or clotting disorder;
* 5.Postoperative complications such as bleeding, pancreatic fistula, gastric obstruction, abdominal infection, and biliary fistula, which made the patient unable to receive adjuvant therapy within 12 weeks after surgery;
* 6. Known allergy to prescription or any component of the prescription used in this study;
* 7. Factors that significantly affect oral drug absorption, such as dysphagia, chronic diarrhea, gastrointestinal obstruction, etc;
* 8. Known HIV, or syphilis infection, or active hepatitis (hepatitis B, hepatitis C);
* 9.Other reasons that are not suitable to participate in this study according to the researcher's judgment

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 146 (Estimated)
Dates: Start 2024-05-01 (Estimated); Primary Completion 2027-05-30 (Estimated); Study Completion 2027-05-30 (Estimated)

PRIMARY OUTCOMES:
relapse-free survival (RFS) | Up to 24 months
  The time from the date of surgery to the disease recurrence or death, whichever is earlier.

SECONDARY OUTCOMES:
distant metastasis-free survival (DMFS) | Up to 24 months
  The time from the date of surgery to the first distant metastasis or death due to any cause, whichever is earlier.
overall survival (OS) | Up to 24 months
  The time from the date of surgery to death due to any cause.
tumor-related markers | Up to 24 months
  To explore the influence of tumor-related markers (such as KRAS, EGFR) on prognosis.
adverse events | Up to 30 days after last administration.
  Frequency and severity of adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Jihui Hao, Dr, Study Chair — Tianjin Medical University Cancer Institute and Hospital
Locations (1):
- Tianjin Medical University Cancer Institute and Hospital, Tianjin, China

IPD SHARING:
Plan to Share IPD: No